CLINICAL TRIAL: NCT05452655
Title: Effects of Intensive Multidisciplinary Rehabilitation and Identification of New Biomarkers in Response to an Integrated Motor-Cognitive and Aerobic Exercises Approaches in People With Parkinson's Disease
Brief Title: Intensive Multidisciplinary Rehabilitation and Biomarkers in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11_16/04/2020
Record Dates: First submitted 2022-05-30; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease; Biomarkers; Rehabilitation Outcome; Gait Disorders, Neurologic; Parkinsonian Disorders; Basal Ganglia Diseases; Central Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases; Cognitive Impairment; Gait Analysis; Pathologic Processes; Magnetic Resonance Imaging; Physiotherapy
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic; Parkinsonian Disorders; Basal Ganglia Diseases; Central Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases; Cognitive Dysfunction; Pathologic Processes

STUDY DESIGN:
Intervention Model Description: This study is designed as a Randomized Controlled Trial (RCT). Subjects with a diagnosis of PD in accordance of MDS criteria will be randomly allocated to the experimental (EXP) or control group (CTR).
  Clinical, kinematic, blood samples and MRI data will be collected before (T0) at the end of treatment (T1) and 3 months after the end of treatment (T2).
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Outpatient Integrated Motor-Cognitive and Aerobic Exercises Rehabilitation Program (Experimental): Intervention of highly challenging motor and cognitive training for 6 consecutive weeks.
  Interventions: Behavioral: Multidisciplinary Intensive Rehabilitation
- Home-Based Stretching Exercises (Active Comparator): Home-based self-treatment program for 40 '/ day for 6 consecutive weeks
  Interventions: Behavioral: Muscle-stretching and active mobilization exercises

INTERVENTIONS:
Behavioral: Multidisciplinary Intensive Rehabilitation — The rehabilitation program will last for 6 consecutive weeks and involves the execution of 30 sessions, 5 days a week lasting 160 '/ day each (80' motor; 40 'cognitive and 40' speech therapy rehabilitation) for 3 days a week and 180'/ day (80 'motor; 60' cognitive and 40 'speech therapy rehabilitation) for 2 days a week. The EXP group will receive 18 sessions (3 times a week) of treadmill (20 min), balance exercises and functional reinforcement (20 min). The remaining motor sessions will be defined based on the patient's therapeutic needs.
  The cognitive treatment will be proposed both in traditional mode (3 times a week) and through the support of semi-immersive "Virtual Reality Rehabilitation System" (VRRS) (2 times/week). The VRRS treatment is structured in 2 sessions per week (60 min) for 6 consecutive weeks.
  The speech therapy program will include clinical and instrumental evaluations and innovative techniques will be used for the treatment (biofeedback with Vitalstim).
  Arms: Intensive Outpatient Integrated Motor-Cognitive and Aerobic Exercises Rehabilitation Program
Behavioral: Muscle-stretching and active mobilization exercises — The control group subjects will undergo a home-based self-treatment program for 40 '/ day for 6 consecutive weeks consisting of muscle-stretching and active mobilization exercises.
  Arms: Home-Based Stretching Exercises

SUMMARY:
Parkinson's disease (PD) is a progressive neurological disorder characterized by motor and non-motor symptoms such as rigidity, bradykinesia, resting tremor, cognitive and autonomic dysfunctions, gait and balance difficulties.

The impairment of gait, balance and cognitive performances is partially responsive to dopaminergic medications. This emphasizes the importance of non-pharmacological interventions for people with PD (pwPD).

Intensive multidisciplinary motor and cognitive rehabilitation has been proposed as a complementary and effective treatment for managing pwPD.

Several structural and physiological mechanisms have been suggested to underpin exercise-induced neuroplastic changes in PD, such as enhanced synaptic strength and preservation of dopamine neurons. To date, studies on brain changes induced by motor and cognitive exercises in pwPD have been small-scaled and uncontrolled.

Identifying accessible and measurable biomarkers for monitoring the events induced by intensive motor and cognitive rehabilitation program would help in testing the treatment effectiveness and would allow personalization of rehabilitation strategies by predicting patients' responsiveness.

Based on validated clinical assessments of intensive multidisciplinary rehabilitation treatment, the project will test the ability of a new set of biomarkers to evaluate rehabilitative outcomes in a cohort of people with PD.

DETAILED DESCRIPTION:
While pharmacological treatment is helpful in the early stages of the disease, increased attention has been given to rehabilitation that may lead to clinical improvements in motor and non-motor impairments.

Recently synthesized evidence suggests that physical exercise may lead to neuroplastic changes at the functional, structural and molecular levels.

Accessible and measurable biomarkers are needed to monitor the disease progression and the neurobiological changes resulting from pharmacological and rehabilitative treatments, also can be a useful and valuable tool to test rehabilitation effectiveness.

The present project will start from the reliable clinical assessment of rehabilitation effectiveness of an intensive multidisciplinary rehabilitation program, to verify the ability of a new panel of measurable biomarkers to assess neurobiological and functional changes in pwPD.

The purpose of this study is to determine the effects of an intensive multidisciplinary, aerobic, motor-cognitive rehabilitation treatment on accessible and measurable molecular biomarkers (primary outcome); balance and gait performance; aerobic capacity; motor and non-motor symptoms; cognitive functions; neuroimaging biomarker (secondary outcomes) in comparison to an active control group receiving a home-based self-treatment program. Thereafter, the investigators aim to relate the effects seen in motor and "non-motor" behavior to changes in biomolecular and neuroimaging markers.

To achieve this purpose, the study is designed as a Randomized Controlled Trial (RCT) and participants will be recruited at Fondazione Don C. Gnocchi-ONLUS, IRCCS S. Maria Nascente. Seventy-two subjects with a diagnosis of PD in accordance of MDS criteria will be randomly allocated to the experimental (EXP) or control group (CTR).

ELIGIBILITY:
Inclusion Criteria:

* PD diagnosis according to MDS Criteria (MDS clinical diagnostic criteria for Parkinson's disease, Postuma et al., 2015);
* Modified Hoehn&Yahr (H&Y): stages from 1.5 to- 3;
* Stable pharmacological treatment in the last 4 weeks.

Exclusion Criteria:

* Vascular, familiar and drug- induced forms of parkinsonism, other known or suspected causes of parkinsonism (metabolic, brain tumor etc) or any suggestive features of atypical parkinsonism;
* Significant comorbidities and/or severe systemic diseases that would preclude exercise participation (eg.recent surgery, unstable cardiac dysfunction, anemia, hepatosis, pulmonary disorders, chronic renal failure; auditory, visual and/or vestibular dysfunctions, presence of DBS); previously diagnosed psychiatric diseases.
* Dementia as defined by Montreal Cognitive Assessment (MoCA Test) Correct Score<15.51 (Santangelo et al., 2014);
* Rehabilitation treatment in the previous 4 weeks.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Serum biomarkers in neuron derived extracellular vesicles (NDEVs) | 18 weeks
  Oligomeric α-synuclein (α-syn) ng/ml; SNARE complex: Syntaxyn-1(STX-1A) (ng/ml), VAMP-2 (ng/ml) and SNAP-25 (ng/ml); Brain-Derived Neurotrophic Factor (BDNF) (ng/ml), pro-BDNF (ng/ml), Glial cell line-derived Neurotrophic factor (GDNF) (ng/ml) Cerebral dopamine neurotrophic factor (CDNF) (ng/ml)
Blood Biomarkers | 18 weeks
  Pro- [IL-1β (pg/ml), Tumour Necrosis Factor alpha (TNFα) (pg/ml), Interferon gamma (IFN-γ) (pg/ml), IL-6 (pg/ml), IL-18 (pg/ml)], Anti-inflammatory (IL-10) (pg/ml) cytokines.

SECONDARY OUTCOMES:
Dynamic Balance | 18 weeks
  - Timed-Up and -Go Test (TUG); subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again. The Time (seconds) is measured.
Aerobic capacity and endurance | 18 weeks
  6 Minute Walk Test (6-MWT). The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Gait speed | 18 weeks
  10 Meter Walk Test (10MWT) assess walking speed in meters per second over a distance of 6 meters.
Strenght | 18 weeks
  5-Time Sit-To-Stand (5TSTS) is based on the amount of time (in seconds) a patient is able to transfer from a seated to a standing position and back to sitting five times.
Balance | 18 weeks
  Modified Dynamic Gait Index (mDGI): The mDGI measure balance skills consists of 8 items and results in a total score of 0 to 64.
Gait Analysis | 18 weeks
  Gait analysis will be assessed using a 9-camera SMART-D motion capture system (BTS, Milano, Italy) in order to measure stride length, step width and length, kinematic data and energy recovery.
Motor and non-motor symptoms | 18 weeks
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I-IV.
  MDS-UPDRS-PART I ''nonmotor experiences of daily living -nM-EDL-" range: 0-52, 0=better outcome, 52=worse outcome; PART-II ''motor experiences of daily living -M-EDL-'' range: 0-52, 0=better outcome, 52=worse outcome; PART-III ''motor examination'' range: 0-132, 0=better outcome, 132=worse outcome; PART IV ''motor complications'' range: 0-24, 0=better outcome, 24=worse outcome.
Non-Motor symptoms | 18 weeks
  Non-Motor Symptoms Scale (NMSS) [range: 0-360, 0=better outcome, 360=worse outcome];
Fatigue | 18 weeks
  Parkinson Fatigue Scale (PFS) [range: 1-5, 1=better outcome, 5=worse outcome];
Daytime sleepiness | 18 weeks
  Epworth Sleepiness Scale (ESS) [range: 0-24, 0=better outcome, 24=worse outcome];
Sleep quality | 18 weeks
  Pittsburgh Sleep Quality Index (PSQI) [range: 0-21, 0=better outcome, 21=worse outcome];
Rapid eye movement sleep behavior disorder | 18 weeks
  REM sleep behavior disorder screening questionnaire (RBDSQ) [range: 0-13, 0=better outcome, 13=worse outcome].
Autonomic Symptoms | 18 weeks
  Italian version of the Composite Autonomic Symptoms Score (COMPASS-31) [weighted score range: 0-100, 0=better outcome, 100=worse outcome];
Pain Intensity | 18 weeks
  Numeric Rating Scale (NRS) [range: 0-10, 0=better outcome, 10=worse outcome];
Parkinson's disease-specific health related quality of life | 18 weeks
  The Parkinson Disease Questionnaire (PDQ-39) [PDQ-39 range: 0%-100%; 0%=better outcome, 100%=worse outcome].
Global Cognitive Functioning | 18 weeks
  Montreal Cognitive Assessment (MoCA Test)[0-30, 0=worse, 30=better outcome] and Mini-Mental Parkinson (MMP)[0-32, 0=worse, 32=better outcome]
Verbal short-term and working memory | 18 weeks
  Forward and Backward Verbal Span [0-9, 0=worse, 9=better outcome]
Verbal episodic memory | 18 weeks
  Immediate and delayed story recall test [0-8, 0=worse, 8=better outcome; Oblivion Index range: 0-8, 0=worse, 8=better outcome]
Visuo-constructional ability | 18 weeks
  Rey's Figure - Copy [0-36, 0=worse, 36=better outcome]
Visuo-spatial memory | 18 weeks
  Rey's Figure - Recall [0-36, 0=worse, 36=better outcome]
Frontal lobe functioning | 18 weeks
  Frontal Assessment Battery (FAB) [0-18, 0=worse, 18=better outcome]
Non-verbal reasoning | 18 weeks
  Raven Coloured Progressive Matrices (CPM-47) [0-36, 0=worse, 36=better outcome]
Extradimensional verbal set-shifting | 18 weeks
  Alternate Verbal Fluency [0-∞, 0=worse, ∞=better outcome;Shifting Index 0-1, 0=worse, 1=better outcome]
Extradimensional non-verbal set-shifting | 18 weeks
  Trail Making Test (TMT) [0-∞, 0=worse, ∞=better outcome]
Speed information processing | 18 weeks
  Symbol Digit Modalities Test (SDMT) (Oral Version) [0-120, 0=worse, 120=better outcome]
Cognitive interference inhibition | 18 weeks
  Stroop Test-Short Version [Error: 0-30, 0=better, 30=worse outcome;Time: range: 0-∞, 0=better, ∞=worse outcome]
IdeoMotor praxis | 18 weeks
  Gesture Imitation Test (IMA-T) [0-72, 0=worse, 72=better outcome]
Language production and non-motor processing speed | 18 weeks
  Verbal fluency test (phonemic and semantic tasks) [0-∞, 0=worse, ∞=better outcome]
Depression | 18 weeks
  Beck Depression Inventory-II (BDI-II) [0-63, 0=better, 63=worse outcome]
Anxiety | 18 weeks
  State-Trait Anxiety Inventory. Forma Y (STAI-Y) [20-80; STAI-Y TRAIT ANXIETY range: 20-80; 20=better, 80=worse outcome]
Apathy | 18 weeks
  Dimensional Apathy Scale (I-DAS) [0-72, 0=better, 72=worse outcome]
Anhedonia | 18 weeks
  Snaith-Hamilton Pleasure Scale (SHAPS) [0-14, 0=better, 14=worse outcome]
Impulsivity | 18 weeks
  Barratt Impulsiveness Scale-11 (BIS-11) [30-120, ;30=better, 120=worse outcome]
Alexithymia | 18 weeks
  Toronto Alexithymia Scale (TAS-20) [20-100, 20=better, 100=worse outcome]
Impulsive Control Disorders | 18 weeks
  Questionnaire for Impulsive-Compulsive Disorders in Parkinson's disease (QUIP-RS-IT) [0-112,; 0=better, 112=worse outcome]
Behavioral disturbances | 18 weeks
  NeuroPsychiatric Inventory Questionnaire (NPI-Q) [SE: 0-36, 0=better, 36=worse outcome; ST= 0-60, 0=better, 60=worse outcome]
Functional disability | 18 weeks
  Modified Barthel Index (MBI) [range: 0-100, 0=worse outcome, 100=better outcome];
Daily self-care activities | 18 weeks
  Activities of Daily Living (ADL) [0-6, 0=worse, 6=better outcome] Instrumental Activities Of Daily Living (IADL) [0-8, 0=worse, 8=better outcome]
Caregiver burden | 18 weeks
  Caregiver Burden Inventory (CBI) [range 0-96, 0=better, 96=worse outcome]
Brain functional connectivity | 18 weeks
  Advanced Magnetic Resonance Imaging (MRI)-3 Tesla protocols, including resting state functional MRI to assess the neural correlates of rehabilitation-induced brain plasticity in pwPD undergoing intensive motor and cognitive rehabilitation.
Cerebral blood flow | 18 weeks
  Advanced MRI-3 Tesla protocols, including arterial spin labeling (ASL) to assess the neural correlates of rehabilitation-induced brain plasticity in pwPD undergoing intensive motor and cognitive rehabilitation.
Home-based motor activity monitoring | 18 weeks
  The acquisitions will be obtained from the actigraphs (mounted one on the right wrist and the other on the left wrist).

CONTACTS AND LOCATIONS:
Overall Officials: Mario Meloni, MD;PhD, Principal Investigator — IRCCS S. Maria Nascente, Fondazione Don Carlo Gnocchi ONLUS
Locations (1):
- IRCCS S. Maria Nascente, Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saibene FL, Agliardi C, Salvatore A, Arcuri P, Castagna A, Gobbo S, Merlo F, Bowman T, Anastasi D, Pagliari C, Farina E, Alberoni M, Calabrese E, La Rosa F, Arienti C, Saresella M, Guerini FR, Cattaneo D, Baglio F, Clerici M, Navarro J, Meloni M. Investigating the effects of a daily multidisciplinary intensive outpatient rehabilitation program on innovative biomarkers in people with Parkinson's disease: Study protocol for a phase III randomized controlled clinical trial. PLoS One. 2024 Oct 23;19(10):e0309405. doi: 10.1371/journal.pone.0309405. eCollection 2024. PMID 39441873